CLINICAL TRIAL: NCT06868693
Title: Pancreatic Cancer of the Head: Effect of Neoadjuvant Chemotherapy in Elderly People - a Multicenter Observational Study
Brief Title: Neoadjuvant Chemotherapy for Elderly with Pancreatic Head Cancer
Acronym: PEACE
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Elena Orlandi, MD (Doctor of Medicine), Azienda Unita Sanitaria Locale di Piacenza
Other Study IDs: PEACE
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer Resectable; Pancreatic Cancer Stage II; Neoadjuvant Therapy; Elderly; Borderline Pancreatic Inoperable Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Neoadjuvant Therapy; N-acetyltalosaminuronic acid; Population Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upfront Surgery (UFS) Group: This cohort includes elderly patients (≥70 years) with resectable or borderline resectable (BR) pancreatic ductal adenocarcinoma (PDAC) who underwent upfront surgical resection (pancreaticoduodenectomy) without prior neoadjuvant therapy. The study will compare oncologic outcomes, including OS, PFS, R0 resection rates, and postoperative complications, between patients receiving NAT and those undergoing immediate surgery.
  Interventions: Drug: Neoadjuvant Chemotherapy (NAT) Group

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy (NAT) Group — This cohort includes elderly patients (≥70 years) with resectable or borderline resectable (BR) pancreatic ductal adenocarcinoma (PDAC) who underwent neoadjuvant chemotherapy (NAT). The NAT regimens include 5-FluoroUracil, Irinotecan, Oxaliplatin (FOLFIRINOX), gemcitabine/nab-paclitaxel (GnP), and other standard chemotherapy protocols. The study aims to evaluate the impact of NAT on overall survival (OS), progression-free survival (PFS), R0 resection rates, and postoperative outcomes, as well as the toxicity profile of different NAT regimens.

SUMMARY:
The goal of this observational retrospective cohort study is to evaluate the efficacy and safety of neoadjuvant chemotherapy (NAT) in elderly patients with resectable or borderline resectable (BR) pancreatic ductal adenocarcinoma (PDAC). The study includes patients aged ≥70 years who have undergone NAT followed by surgery or upfront surgery.

The main questions it aims to answer are:

Does NAT improve overall survival (OS) and progression-free survival (PFS) in elderly patients compared to upfront surgery? What is the impact of NAT on R0 resection rates, conversion rates in BR tumors, and the need for vascular resection? How does the toxicity profile of different NAT regimens affect treatment outcomes and patient tolerability? Researchers will compare NAT followed by surgery vs. upfront surgery to determine differences in oncologic outcomes and postoperative complications.

Participants will:

Be retrospectively identified from hospital records. Be classified based on treatment received (NAT vs. upfront surgery). Undergo data collection on tumor characteristics, treatment regimens, surgical details, and survival outcomes.

This study aims to refine patient selection criteria for NAT in elderly patients, guiding personalized treatment strategies to optimize survival and quality of life.

ELIGIBILITY:
Inclusion Criteria

* Patients aged ≥ 70 years
* Patients with resectable or BR PDAC who underwent curative treatment (NAT followed by surgery and upfront surgery)
* Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) > 2
* Patients able to provide informed consent, whenever possible

Exclusion Criteria

* Patients not meeting the inclusion criteria.
* Pancreatic cancer of pancreatic body and tail.
* Patients with metastatic disease.
* Patients with locally advanced or metastatic pancreatic cancer

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of elderly patients (≥70 years old) diagnosed with resectable or borderline resectable (BR) pancreatic ductal adenocarcinoma (PDAC). Patients will be retrospectively identified from hospital databases and electronic medical records across multiple international and multicenter institutions.
  Participants included in the study have undergone either neoadjuvant chemotherapy (NAT) followed by surgery or upfront surgery (pancreaticoduodenectomy). Data will be collected from oncology, surgery, and gastroenterology units within tertiary referral centers and high-volume pancreatic cancer treatment centers.
  The study focuses on real-world clinical practice and aims to evaluate treatment outcomes, including overall survival, disease progression, surgical resection rates, and treatment-related toxicities, in this clinically vulnerable population.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 2 years from treatment initiation
  OS is defined as the time from the initiation of treatment (NAT or upfront surgery) to death from any cause. Patients still alive at the end of the study period will be censored at the last follow-up date.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 1 years from treatment initiation
  PFS is defined as the time from the initiation of treatment to disease progression or death from any cause, whichever occurs first. Disease progression is assessed based on RECIST v1.1 criteria using imaging studies.
Resection Rate and R0 Resection Rate | At the time of surgery
  The proportion of patients who successfully undergo surgical resection after NAT compared to upfront surgery. Resection margins will be classified as:
  R0 (complete resection, negative margins) R1 (microscopic residual disease) R2 (macroscopic residual disease)
Major Toxicities and NAT Dropout Rate | At the end of each cycle (each cycle is 28 days)
  Toxicity will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. The study will report grade 3-4 toxicities, dose reductions, treatment interruptions, and patient dropout rates due to adverse events.
Conversion Rate of NAT in Borderline Resectable (BR) PDAC | At the time of surgery
  The proportion of patients initially classified as borderline resectable (BR) who are successfully converted to resectable status after NAT and undergo curative-intent surgery.
Vascular Resection Rate | At the time of surgery
  Comparison of the frequency of vascular resections (e.g., portal vein or superior mesenteric vein resection) between the NAT and upfront surgery groups, assessing the impact of NAT on vascular involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Giuffrida, MD, Principal Investigator — AUSL Piacenza; Elena Orlandi, MD, Principal Investigator — AUSL Piacenza

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR